CLINICAL TRIAL: NCT03493737
Title: Cost-Utility Evaluation Comparing Hospital Versus Home-Based Bortezomib in Multiple Myeloma: The ADHOMY Study
Brief Title: Cost-Utility Analysis Hospital Versus Home in Multiple Myeloma
Acronym: ADHOMY
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A00103-52
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HaH (Hospital-at-Home): Bortezomib is injected at Outpatient hospital at day 1 and at Home at further day of cycles
  Interventions: Behavioral: Quality of life surveys
- OH (Outpatient Hospital): Bortezomib is always injected at Outpatient hospital
  Interventions: Behavioral: Quality of life surveys

INTERVENTIONS:
Behavioral: Quality of life surveys — Quality of life surveys by EQ-5D and QLQ-C30

SUMMARY:
Bortezomib needs repetitive visits at hospital for injections. Hospital-at-Home (HaH) might be an attractive and suitable alternative in this situation.

This study aim to perform a cost-utility analysis of two different strategies in several HaH structures within the Grand Est region in France.

DETAILED DESCRIPTION:
Bortezomib is a standard therapy of newly-diagnosed multiple myeloma and is also approved for relapsing disease, requiring the patients to travel to the outpatient-hospital (OH) once a week for several months. Hospital-at-Home (HaH) might be an attractive and suitable alternative in this situation.

This study aim to perform a cost-utility analysis of two different strategies in several HaH structures within the Grand Est region in France: exclusive hospital-based Bortezomib administration versus combined administration in both OH and HaH.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 18
* Enrolled in a social security scheme
* Diagnosis of multiple myeloma in first line or relapse
* Treatment plan including Bortezomib, adopted in a multidisciplinary meeting in a department of Hematology in Nancy (main investigator), Reims, Strasbourg University Hospitals or Metz-Thionville and Mulhouse local state-run hospitals
* The patients must have agreed to the treatment protocol and to take IV or PO associated drugs prescribed in addition to Bortezomib
* The patients must meet the 2003 eligibility criteria of the National Agency for Accreditation and Evaluation in Health (ANAES) for chemotherapy at home:

  * Absence of severe adaptive or psychological disorders, ability to understand the protocol
  * Absence of cognitive impairment
  * Availability and agreement of the attending physician
  * Home safety and hygiene
* Do not decline to participate in the research and share their personal data

Exclusion Criteria:

* Already participating in another trial
* Have a follow-up and/or treatment for another condition requiring a particular care during the Bortezomib treatment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple myeloma requiring a treatment with Bortezomib
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Cost therapy assessment | 10 months follow-up per patient
  Cost therapy assessment including direct medical costs, non-medical costs and indirect costs, investigated from the French Health Insurance perspective and expressed in Euro.
EQ-5D questionnaire | 10 months follow-up per patient
QLQ-C30 questionnaire | 10 months follow-up per patient
  an oncology-specific instrument

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided